CLINICAL TRIAL: NCT05140759
Title: A Multi-centre, Prospective, Open Label, Uncontrolled Pilot Study to Assess the Feasibility and Tolerability of an Automated Continual Water Removal System in Patients With Advanced Diuretic Resistant Heart Failure
Brief Title: An Automated Continual Water Removal System in Patients With Advanced Diuretic Resistant Heart Failure
Acronym: ACWR-HF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: challenges in recruitment
Sponsor: Paragate Medical LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PM-2020-10000 IPUDX
Record Dates: First submitted 2021-11-09; First posted 2021-12-01 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Implanted device (Experimental): Implantation and activation of an automated continual water removal system, including 4-months follow up
  Interventions: Device: automated continual water removal system

INTERVENTIONS:
Device: automated continual water removal system — The device removes excess fluids in heart failure patients with diuretic resistance

SUMMARY:
This study will assess the functionality and tolerability of an automated continual water removal system in up to 8 patients with HF and diuretic resistance.

intervention: Implanted absorption chamber, connected to an external pump. Follow up: 3 months post activation.

DETAILED DESCRIPTION:
Study Duration: 24 months Enrolment 20 months, Follow-up 3 months, Close-out 1 month Study Centres Up to 4 centres with Medical University Wroclaw, Poland, as the principal site.

Objectives: To assess the feasibility, tolerability and functionality of an intra-peritoneal, mechanically induced, ultrafiltration system, through the analysis of procedure and device related serious adverse events and device function.

Number of Subjects: Up to 8 Diagnosis and Main Inclusion Criteria: Patients with fluid overloaded congested heart failure (NYHA Class II-IV) with diuretic resistance and a history of multiple heart failure related admissions.

Study Product and Planned Use: The Paragate Medical IPUDx System comprises an intraperitoneally implanted fluid absorption chamber with an external wearable rechargeable pump, drainage bag and controller. The system induces isotonic fluid loss across the peritoneal membranes which is collected in the fluid absorption chamber and transported to the external fluid drainage bag.

Statistical Methodology: No statistical hypothesis is proposed. Safety will be evaluated using a complete description of Serious Adverse Events. A descriptive analysis will be performed for all primary and secondary variables of the study for the basal measures and all post-basal measures.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 21 years of age

  * Life expectancy > 6 months
  * HF, NYHA class II-IV
  * > 1 HF related admissions in the last 12 months
  * Fluid congestion (2 signs of pitting oedema, jugular distention, BW elevation, nocturnal dyspnoea score, respiration rate, pulmonary congestion and/or pleural effusion per chest x-ray, ascites)
  * Failure to achieve effective diuresis and congestion relief despite appropriate or escalating diuretic doses or combination of diuretics (eg. Furosemide and Metolazone)
  * Eligible for general anaesthesia and laparoscopic procedure
  * Able to give written informed consent
  * Ability to comply with study procedures and ability to operate the device
  * Women of childbearing potential should use adequate contraception for as long as the device is implanted.

Exclusion Criteria:

* • Any non-cardiac disease with life expectancy < 1 year

  * Any patient listed for solid organ transplantation
  * Patients with history, or with indication for, mechanical circulatory support
  * iv inotropes required in last 3 months (INTERMACS Score ≤3)
  * Immunocompromised (e.g. chronic steroid treatment, HIV, etc.)
  * Insulin dependent diabetes
  * Severe hyponatraemia as defined by a serum Sodium < 120 mmol/l
  * Serum Albumin < 2.5 g/dL
  * eGFR < 25 ml/min/1.73m2 by MDRD method
  * Previous significant intraabdominal surgery, severe abdominal adhesions, intra-abdominal foreign body (except for small inguinal mesh)
  * Large diaphragmatic hernia, or surgically irreparable, complex or recurring hernia
  * 6 minutes' walk test of less than 100 meter
  * History (>6 months) of diaphragmatic hernia, inflammatory or ischemic bowel disease and frequent episodes of diverticulitis
  * Gastrointestinal haemorrhage within the last 4 months
  * Bacterial peritonitis episode within the last 24 months
  * > 2 systemic or local infections, such as urinary tract infection or abdominal skin infection within the last 6 months
  * Liver cirrhosis
  * BMI > 40 presenting a risk for surgery
  * Patients with contraindications for general anaesthesia or laparoscopic surgery
  * Unsuitability for self-maintenance of the experimental home set-up
  * Presence of any current cancer
  * Presence of any active implantable or body-worn devices that cannot be removed excluding ICD / pacemaker
  * Pregnancy
  * Patients being in another therapeutic clinical study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2024-01-17 (Actual)

PRIMARY OUTCOMES:
Analysis of AEs related to implantation | 4 months
  Analysis of incidence and severity of AEs that occur during or following implantation and are related to it.
Analysis of AEs related to the device and its function. | 4 months
  Analysis of incidence and severity of AEs related to the device and its function.

SECONDARY OUTCOMES:
Functionality | 4 months
  Assessed by a daily volume of fluid removal
Clinical assessment of fluid overload | 4 months
  Fluid retention measures such as pitting oedema, jugular distention, body weight elevation
Echocardiographic assessment of LVESD, LVEDD, and LVEF | 4 months
  Data from echocardiography will enable the provision of volumes, diastolic function, right ventricular function, hemodynamics, and valvular regurgitation.
  This versatile tool is employed vastly for the management of heart failure.
  LVEF - Left Ventricular Ejection Fraction LVESD -Left Ventricular End-Systolic Diameters LVEDD - Left Ventricular external end-diastolic diameter
Quality of life questionnaire | 4 months
  KCCQ-12 questionnaire
  The Kansas City Cardiomyopathy Questionnaire (KCCQ) is a 23-item self-administered questionnaire developed to independently measure the patient's perception of their health status, which includes heart failure symptoms, impact on physical and social function, and how their heart failure impacts their quality of life (QOL) within a 2-week recall period.
  KCCQ scores are scaled from 0 to 100 and frequently summarized in 25-point ranges, where scores represent health status as follows: 0 to 24: very poor to poor; 25 to 49: poor to fair; 50 to 74: fair to good; and 75 to 100: good to excellent.
Nocturnal dyspnea score | 4 months
  Will be assessed using the following questions:
  Has the patient ever woken up at night with shortness of breath? How long after lying down did the episode occur?
  Number of pillows used under the patient's head at night:
  Has the patient ever had to sleep sitting up? Has the patient developed coughing or wheezing in the recumbent position? What did the patient do to relieve his distress? Please specify.
6 minutes' walk test | 4 months
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
NT-proBNP | 4 months
  NT-proBNP is a marker for HF severity.
Serum Creatinine | 4 months
  A marker for kidney function.
Serum / urine electrolytes levels. | 4 months
  Electrolyte and metabolite disorders indicate on kidney function.
  hypercalcemia /hypocalcemia. hyperchloremia /hypochloremia. hypermagnesemia /hypomagnesemia. hyperphosphatemia /hypophosphatemia. hyperkalemia /hypokalemia. hypernatremia /hyponatremia.

CONTACTS AND LOCATIONS:
Overall Officials: Aharon Abbo, MD, Principal Investigator — Rambam Health Care Campus; Robert Zymlinski, MD, Principal Investigator — Uniwersytecki Szpital Kliniczny im Jana Mikulicza-Radeckiego, ul. Borowska 213, 50-556 Wrocław; Paata Meshveliani, MD, Principal Investigator — West Georgian Medical Center
Locations (3):
- West Georgian Medical Center, Kutaisi, Georgia
- Rambam medical center, Haifa, Israel
- Uniwersytecki Szpital Kliniczny im Jana Mikulicza-Radeckiego, Wroclaw, Poland